CLINICAL TRIAL: NCT02902471
Title: Functional Evaluation of Distal Airways by Forced Oscillations: Diagnosis Help in Bronchiolitis Obliterans Syndrome in Post Bone Marrow Transplantation
Brief Title: Forced Oscillations for Diagnosis Help in Bronchiolitis Obliterans Syndrome in Post Bone Marrow Transplantation
Acronym: OSCILLOMOELL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2010/48; 2010-A01229-30 (Other: ANSM)
Record Dates: First submitted 2016-09-12; First posted 2016-09-15 (Estimated); Last update posted 2018-07-16 (Actual); Status verified 2017-04

CONDITIONS: Bronchiolitis Obliterans; Bone Marrow Transplantation
MeSH Terms: conditions — Bronchiolitis Obliterans

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Group A (Experimental): Patients with bronchiolitis obliterans syndrome after bone marrow transplantation
  Interventions: Other: Forced oscillations measure

INTERVENTIONS:
Other: Forced oscillations measure

SUMMARY:
A study to evaluate the role of forced oscillations in diagnosis of bronchiolitis obliterans syndrome in patients after bone marrow transplantation. The force oscillations technique will be compared with classical spirometry.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years
* Bone marrow or hematopoietic stem cells transplantation for more than 100 days
* Clinical stability
* Patients affiliated to a social security system
* Patients having given his (her) written consent.

Exclusion Criteria:

* Bronchiolitis Obliterans already diagnosed
* Unresolved Respiratory infection
* Unresolved mechanical complication (pneumothorax, effusions)
* Medicinal pneumopathy
* Inability to perform pulmonary function tests

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2011-06; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Number of days | 2 years
  Temporal difference between the date of the functional change measured by the technique of the forced oscillations and by the standard techniques of plethysmography.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Louis Couderc, MD, PhD, Principal Investigator — Hopital Foch
Locations (2):
- France (2):
  - CHRU de Lille, Lille
  - Hopital Foch, Suresnes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Williams KM, Chien JW, Gladwin MT, Pavletic SZ. Bronchiolitis obliterans after allogeneic hematopoietic stem cell transplantation. JAMA. 2009 Jul 15;302(3):306-14. doi: 10.1001/jama.2009.1018. PMID 19602690
- [Background] Soubani AO, Uberti JP. Bronchiolitis obliterans following haematopoietic stem cell transplantation. Eur Respir J. 2007 May;29(5):1007-19. doi: 10.1183/09031936.00052806. PMID 17470622
- [Background] Chien JW, Martin PJ, Gooley TA, Flowers ME, Heckbert SR, Nichols WG, Clark JG. Airflow obstruction after myeloablative allogeneic hematopoietic stem cell transplantation. Am J Respir Crit Care Med. 2003 Jul 15;168(2):208-14. doi: 10.1164/rccm.200212-1468OC. Epub 2003 Mar 20. PMID 12649126
- [Background] Bergeron A, Belle A, Chevret S, Ribaud P, Devergie A, Esperou H, Ades L, Gluckman E, Socie G, Tazi A. Combined inhaled steroids and bronchodilatators in obstructive airway disease after allogeneic stem cell transplantation. Bone Marrow Transplant. 2007 May;39(9):547-53. doi: 10.1038/sj.bmt.1705637. Epub 2007 Mar 12. PMID 17351647
- [Background] Gunn ML, Godwin JD, Kanne JP, Flowers ME, Chien JW. High-resolution CT findings of bronchiolitis obliterans syndrome after hematopoietic stem cell transplantation. J Thorac Imaging. 2008 Nov;23(4):244-50. doi: 10.1097/RTI.0b013e3181809df0. PMID 19204468
- [Background] Martin PJ, Weisdorf D, Przepiorka D, Hirschfeld S, Farrell A, Rizzo JD, Foley R, Socie G, Carter S, Couriel D, Schultz KR, Flowers ME, Filipovich AH, Saliba R, Vogelsang GB, Pavletic SZ, Lee SJ; Design of Clinical Trials Working Group. National Institutes of Health Consensus Development Project on Criteria for Clinical Trials in Chronic Graft-versus-Host Disease: VI. Design of Clinical Trials Working Group report. Biol Blood Marrow Transplant. 2006 May;12(5):491-505. doi: 10.1016/j.bbmt.2006.03.004. PMID 16635784
- [Background] Garcia G, Perez T, Mahut B. [Lung function testing and assessment of distal airways in asthma]. Rev Mal Respir. 2009 Apr;26(4):395-406; quiz 479, 482. doi: 10.1016/s0761-8425(09)74044-6. French. PMID 19421092
- [Background] Bourdin A, Paganin F, Prefaut C, Kieseler D, Godard P, Chanez P. Nitrogen washout slope in poorly controlled asthma. Allergy. 2006 Jan;61(1):85-9. doi: 10.1111/j.1398-9995.2006.00970.x. PMID 16364161
- [Background] Oostveen E, MacLeod D, Lorino H, Farre R, Hantos Z, Desager K, Marchal F; ERS Task Force on Respiratory Impedance Measurements. The forced oscillation technique in clinical practice: methodology, recommendations and future developments. Eur Respir J. 2003 Dec;22(6):1026-41. doi: 10.1183/09031936.03.00089403. PMID 14680096
- [Background] Smith HJ, Reinhold P, Goldman MD. Forced Oscillation Technique and Impulse Oscillometry. Lung Function Testing: European Respiratory Society Monograph. Sheffield, England: European Respiratory Society; 2005:72-105
- [Background] Goldman MD. Clinical application of forced oscillation. Pulm Pharmacol Ther. 2001;14(5):341-50. doi: 10.1006/pupt.2001.0310. PMID 11603948
- [Background] Hamakawa H, Sakai H, Takahashi A, Zhang J, Okamoto T, Satoda N, Aoyama A, Chen F, Fujinaga T, Shoji T, Bando T, Mishima M, Wada H, Date H. Forced oscillation technique as a non-invasive assessment for lung transplant recipients. Adv Exp Med Biol. 2010;662:293-8. doi: 10.1007/978-1-4419-1241-1_42. PMID 20204806
- [Background] Faria AC, Lopes AJ, Jansen JM, Melo PL. Evaluating the forced oscillation technique in the detection of early smoking-induced respiratory changes. Biomed Eng Online. 2009 Sep 25;8:22. doi: 10.1186/1475-925X-8-22. PMID 19781078
- [Background] Brochard L, Pelle G, de Palmas J, Brochard P, Carre A, Lorino H, Harf A. Density and frequency dependence of resistance in early airway obstruction. Am Rev Respir Dis. 1987 Mar;135(3):579-84. doi: 10.1164/arrd.1987.135.3.579. PMID 3826883
- [Background] Skloot G, Goldman M, Fischler D, Goldman C, Schechter C, Levin S, Teirstein A. Respiratory symptoms and physiologic assessment of ironworkers at the World Trade Center disaster site. Chest. 2004 Apr;125(4):1248-55. doi: 10.1378/chest.125.4.1248. PMID 15078731
- [Background] Di Mango AM, Lopes AJ, Jansen JM, Melo PL. Changes in respiratory mechanics with increasing degrees of airway obstruction in COPD: detection by forced oscillation technique. Respir Med. 2006 Mar;100(3):399-410. doi: 10.1016/j.rmed.2005.07.005. Epub 2005 Aug 22. PMID 16115754
- [Background] Kanda S, Fujimoto K, Komatsu Y, Yasuo M, Hanaoka M, Kubo K. Evaluation of respiratory impedance in asthma and COPD by an impulse oscillation system. Intern Med. 2010;49(1):23-30. doi: 10.2169/internalmedicine.49.2191. Epub 2010 Jan 1. PMID 20045997
- [Background] Cavalcanti JV, Lopes AJ, Jansen JM, Melo PL. Detection of changes in respiratory mechanics due to increasing degrees of airway obstruction in asthma by the forced oscillation technique. Respir Med. 2006 Dec;100(12):2207-19. doi: 10.1016/j.rmed.2006.03.009. Epub 2006 May 18. PMID 16713226
- [Background] Kim CW, Kim JS, Park JW, Hong CS. Clinical applications of forced oscillation techniques (FOT) in patients with bronchial asthma. Korean J Intern Med. 2001 Jun;16(2):80-6. doi: 10.3904/kjim.2001.16.2.80. PMID 11590906
- [Background] Kolsum U, Borrill Z, Roy K, Starkey C, Vestbo J, Houghton C, Singh D. Impulse oscillometry in COPD: identification of measurements related to airway obstruction, airway conductance and lung volumes. Respir Med. 2009 Jan;103(1):136-43. doi: 10.1016/j.rmed.2008.07.014. Epub 2008 Aug 28. PMID 18760576